CLINICAL TRIAL: NCT00000262
Title: Effects of Combined Sevoflurane and Nitrous Oxide Inhalation
Brief Title: Effects of Combined Sevoflurane and Nitrous Oxide Inhalation - 14
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-08391-14; R01DA008391 (NIH); R01-08391-14
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: nitrous oxide; sevoflurane; drug interaction; subjective effects; analgesia; healthy volunteers
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Agnosia | interventions — Nitrous Oxide; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (3):
- Placebo +/- 30% Nitrous oxide (Placebo Comparator)
  Interventions: Drug: 30% Nitrous oxide; Other: Placebo
- Sevoflurane 0.2% +/- 30% Nitrous oxide (Active Comparator)
  Interventions: Drug: 30% Nitrous oxide; Drug: 0.2% sevoflurane
- Sevoflurane 0.4% +/- 30% Nitrous oxide (Active Comparator)
  Interventions: Drug: 30% Nitrous oxide; Drug: 0.4% Sevoflurane

INTERVENTIONS:
Drug: 30% Nitrous oxide
Drug: 0.4% Sevoflurane
  Arms: Sevoflurane 0.4% +/- 30% Nitrous oxide
Drug: 0.2% sevoflurane
  Arms: Sevoflurane 0.2% +/- 30% Nitrous oxide
Other: Placebo
  Arms: Placebo +/- 30% Nitrous oxide

SUMMARY:
The purpose of this study is to determine the effects of combined sevoflurane and nitrous oxide inhalation on mood, psychomotor performance, and the pain response in humans.

ELIGIBILITY:
Please contact site for information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1996-11; Primary Completion 1999-02 (Actual); Study Completion 1999-02 (Actual)

PRIMARY OUTCOMES:
Pain intensity, pain bothersomeness | During inhalation
  Inhalation was for 68 min divided into 4 blocks with nitrous oxide added during either block 2 or block 4
Mood | During inhalation
  Inhalation was for 68 min divided into 4 blocks with nitrous oxide added during either block 2 or block 4
Psychomotor performance | During inhalation
  Inhalation was for 68 min divided into 4 blocks with nitrous oxide added during either block 2 or block 4

CONTACTS AND LOCATIONS:
Overall Officials: James Zacny, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Anesthesia & Critical Care, Chicago, Illinois, United States